CLINICAL TRIAL: NCT02000401
Title: To Evaluate the Efficacy, Tolerability, and Safety of Intranasal Ketorolac Tromethamine (Sprix) as an Option for Acute (up to 5 Days) Pain Management Adult Interstitial Cystitis Patients Experiencing a Flare of Pain
Brief Title: Intranasal Ketorolac Tromethamine (Sprix) for Acute Pain of Interstitial Cystitis Flare of Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Citrus Valley Medical Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0703-2012-SPRIX
Record Dates: First submitted 2013-11-19; First posted 2013-12-04 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-11

CONDITIONS: Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Ketorolac Tromethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ketorolac Tromethamine (Other): Ketorolac Tromethamine one 15.75 mg spray in each nostril for a total dose of 31.5 mg which can be repeated every 6-8 hrs. as needed for pain with a maximum daily dose of 126 mg. The treatment may be continued for up to 5 days.
  Interventions: Drug: Ketorolac Tromethamine

INTERVENTIONS:
Drug: Ketorolac Tromethamine
  Other Names: SPRIX

SUMMARY:
Intranasal Ketorolac tromethamine has a potential role as a short term pain management tool for Interstitial Cystitis without the risk and undesirable effects of narcotics.

ELIGIBILITY:
Inclusion Criteria:

1. Female Subject must be between the age eighteen (18) years and sixty four (64)
2. Subject must weigh 110lbs (50kg) or greater
3. Willing and able to provide an informed consent
4. Diagnosed with Interstitial Cystitis/Painful Bladder Syndrome (IC/PBS)
5. Symptoms of IC/PBS that are moderate to severe (intermittent or chronic) for ≥ three (3) months
6. A cystoscopic examination under anesthesia with hydro-distention and photo documentation will have been performed at time of diagnosis with IC. Bladder biopsies will have been performed only if carcinoma is suspected. (see exclusion # 5.2.25 - hydrodistention must be performed greater than four (4) weeks prior to baseline visit) Note: at investigator discretion subject may included with only operative report
7. At screening subject must have a score ≥ four (4) out of ten (10) On Visual Analogue Pain Scale (VAS Pain Scale)
8. Subject must have a score on the O'Leary/Sant scale of at least a five (5) on the symptom index at screening
9. Voids greater than eight (8) in a twenty four (24) hour period
10. Nocturia of at least one (1) time during sleeping period
11. Subject of child-bearing potential must test negative for pregnancy prior to treatment or provide documentation for having undergone the following: hysterectomy or tubal ligation. Subjects who are physiologically capable of becoming pregnant must voluntarily sign a pregnancy waiver included within the informed consent and agree not to become pregnant for the duration of the study and for thirty (30) days following the completion of study. If a subject becomes pregnant during the course of this study, the subject will inform the Principal Investigator within one (1) working day of learning of the pregnancy

Exclusion Criteria:

1. Current treatment with or known allergy or sensitivity to all forms of ketorolac tromethamine, aspirin, other non-steroidal anti-inflammatory drugs (NSAIDs) or Ethylenediaminetetraacetic acid (EDTA) NOTE: if at time of signing consent a subject is receiving a non-steroidal inflammatory drug they may washout for seven days prior to completing the screening visit
2. Subject is currently receiving or having had prior IC/PBS focused therapy on less than three (3) months stable doses. i.e. oral Pentosan Polysulfate(PPS) (Elmiron®), Amitriptyline (Elavil®), oxychlorosene (Clorpactin®), dimethyl sulfoxide (RIMSO 50™), heparin or antihistamine NOTE: Antihistamine is allowable as added treatment during course of study if for treatment of diagnosed nasal/seasonal/environmental allergy (i.e treatment other than IC) , If a subject is receiving intravesical instillations of any kind at least a two day washout must be adhered to before screening is performed. The subject must abstain from any intravesical instillation during the study.
3. Current use of TENS (Transcutaneous Electrical Nerve Stimulation) or Interstim unit
4. Clinically significant urinary tract infection (UTI) NOTE: dipstick urinalysis is done at screening urine culture will be performed if indicated by results of dipstick urinalysis at screening
5. As needed Use of narcotics/opiate within one (1) week prior to the screening visit and entire study participation by self-reporting (Note: once subject has qualified they will be given the option of rescue medication for pain not relieved by the study medication)
6. Use of illegal drugs by self-reporting
7. History of drug or alcohol abuse within five (5) years of screening visit
8. History of suicide attempt or suicidal thoughts by self-reporting within five (5) years of screening visit
9. Any active co-morbid pelvic diagnosis (i.e. endometriosis, Irritable Bowel Syndrome, etc.) for which the subject is unable to distinguish between IC/PBS pain and pain from any other condition as determined by the investigator
10. A diagnosis of a severe neuro-psychiatric disease
11. Subject demonstrates an absence of nocturia
12. Subject's frequency of urination is equal to or less than eight (8) times in a twenty four (24) hour period.
13. Subject's symptoms relieved by antimicrobials, urinary antiseptics, anticholinergics, or antispasmodics.
14. Subject has recurrent bladder or lower urethral calculi (recurrent is defined as > to 3 times in a 12 month period)
15. Subject has active genital herpes with a (3) three month period of the screening visit
16. Subject has uterine, cervical, vaginal, or urethral cancer
17. Subject has been administered cyclophosphamide or any agent that causes chemical cystitis
18. Subject has tubercular cystitis
19. Subject has radiation cystitis
20. Subject has benign or malignant bladder tumor
21. Subject has a positive pathologic vaginal culture within three (3) months of the screening visit
22. Subject has evidence of vesicle ureteral reflux or urethral diverticula
23. Subject has neurogenic bladder dysfunction
24. Subject has a prior urinary diversion
25. Subject who is currently receiving investigational drug(s) or participated in a clinical trial involving investigational drug(s) within thirty (30) day of the screening visit
26. Subject who is pregnant or lactating
27. Subject with history of hydro-distention within four (4) weeks of baseline visit
28. Subject with history of clinically significant cardiovascular disease such as: (chronic stable angina being currently treated with long acting nitrates, chronic stable angina require treatment with short acting nitrates with 90 days of visit 1, angina occurring during sexual intercourse in the last six months, unstable angina within six months of visit 1
29. Resting, sitting blood pressure (BP) > 160mm Hg in systolic pressure or > 100mm Hg is diastolic pressure at screening. If a patient is found to have untreated significant hypertension at screening and antihypertensive treatment is initiated, assessment for study eligibility should be deferred until BP and antihypertensive medication have been stable for at least one month. For patients with previously diagnosed hypertension, antihypertensive medications must be stable for at least one month prior to screening.
30. Subject over sixty four (64) years of age
31. Subject who weighs less than 110lbs (50kg)
32. Subject with history of any clinically significant blood chemistry, renal function or liver abnormality defined as + two (2X) normal values
33. Subject who has history of a bleeding problem or low platelet count
34. Known or suspected cerebrovascular bleeding, hemorrhagic diathesis or incomplete hemostasis, and those at high risk of bleeding, have history of a bleeding problem or low platelet count or coagulation disorder or are on therapy that affects homeostasis
35. Active peptic ulcer disease, recent GI bleeding or perforation, or a history of peptic ulcers or GI bleeding
36. History of asthma, urticaria or other allergic-type reaction after taking aspirin or other non- steroidal inflammatory drugs (NASIDs)
37. Subject who has history of swelling of face, mouth, tongue, lips, gums, neck, or throat (angioedema) or with cardiac decompensation or similar conditions
38. Major surgery scheduled within 3 weeks or screening and for entire participation of study
39. Current exfoliative dermatitis, Stevens-Johnson syndrome or toxic epidermal necrolysis
40. Any condition in the opinion of the investigator that makes the subject unsuitable for study

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Pain Scores on the Visual Analog Scale | 5 days

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Edward L Davis, M.D., Principal Investigator — Citrus Valley Medical Research, Inc.
Locations (1):
- Citrus Valley Medical Research, Inc, Glendora, California, United States